CLINICAL TRIAL: NCT00737282
Title: A Phase III, Open-Label, Parallel, Randomized, Multicenter Study Evaluating the Safety of 25 And 50 mg Proellex® (CDB-4124) in the Treatment of Premenopausal Women With Symptomatic Uterine Fibroids
Brief Title: Multicenter Study Evaluating the Safety of Proellex® in Premenopausal Women With Uterine Fibroids
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Repros stopped study for safety and FDA put study on hold.
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZPU-305
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Uterine Fibroids
Keywords: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 25 mg Proellex (Active Comparator): Proellex 25 mg once daily
  Interventions: Drug: Proellex 25 mg
- Proellex 50 mg (Active Comparator): Proellex 50 mg once daily
  Interventions: Drug: Proellex 50 mg

INTERVENTIONS:
Drug: Proellex 25 mg — One capsule Proellex 25 mg administered as daily oral doses for four (4) consecutive months during each treatment cycle
  Other Names: Telapristone acetate
  Arms: 25 mg Proellex
Drug: Proellex 50 mg — Two capsules Proellex 25 mg administered as daily oral doses for four (4) consecutive months during each treatment cycle
  Other Names: Telapristone acetate
  Arms: Proellex 50 mg

SUMMARY:
The safety of Proellex 25 and 50 mg administered once daily for three treatment cycles (four months each) will be evaluated.

DETAILED DESCRIPTION:
Subjects will be randomized to either Proellex dose, 25 mg or 50 mg, in a 1:1 ratio. Subjects will receive drug for a four (4) month cycle of therapy three (3) times, each treatment cycle being separated by an off-drug interval until menstruation occurs. During the treatment periods, all subjects will be assessed monthly. Subjects will undergo an additional follow-up for 3 months following their last treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* Speak, read and understand English or Spanish;
* Not have undergone hysterectomy, uterine arterial embolization or endometrial ablation therapy (previous myomectomy is acceptable) for any cause and no surgical interventions for uterine fibroids (e.g. hysterectomy, myomectomy, uterine arterial embolization) are planned or anticipated during the study;
* One uterine fibroid must be identifiable and measurable by transvaginal ultrasound;
* Menstrual cycle lasting from 24 to 36 days;
* History of excessive menstrual bleeding;
* Negative urine pregnancy test at screening.

Additional inclusion criteria may apply.

Exclusion Criteria:

* Six months or more (immediately prior to Screening Visit) without a menstrual period;
* Prior hysterectomy;
* Prior bilateral oophorectomy;
* Pregnant or lactating females or women who are attempting or expecting to become pregnant at any time during the study;
* Documented endometriosis, active pelvic inflammatory disease (PID), platelet dysfunction, or Von Willebrand's Disease;
* Any history or diagnosis of gynecological cancer or cervical dysplasia of any grade including atypical squamous cells of undetermined significance (ASCUS) associated with Human Papilloma Virus (HPV);
* Subject with diagnosed or suspected carcinoma of the breast, reproductive organs or any other organ system;
* Subject with known active infection with HIV, Hepatitis A, B or C, Gonorrhea, or Chlamydia or previous history of auto-immune disease or positive serum antinuclear antibodies.

Additional exclusion criteria may apply.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre vanAs, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (25):
- United States (25):
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - AWC Clinical Trials LLC, Little Rock, Arkansas
  - Impact Clinical Trials, Beverly Hills, California
  - Genesis Center for Clinical Research, San Diego, California
  - Physician Care Clinical Research, LLC, Sarasota, Florida
  - Atlanta Women's Research Inst, Atlanta, Georgia
  - Medical Network for Education and Research, Decatur, Georgia
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - York Clinical Consulting, Marrero, Louisiana
  - NECCR Falls River LLC, Fall River, Massachusetts
  - ClinSite, LLC, Ann Arbor, Michigan
  - Female Pelvic Medicine, Grand Rapids, Michigan
  - Alegent Research, Omaha, Nebraska
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - Clinical Trials of America, Eugene, Oregon
  - Thomas Jefferson University - Jefferson Center for Women's Medical Specialties, Philadelphia, Pennsylvania
  - University Medical Group, Dept of OB/GYN, Greenville, South Carolina
  - Greenville Pharmaceutical Research, Greenville, South Carolina
  - Memphis Women's Healthcare, Memphis, Tennessee
  - Women's Care Center, PLC Research Memphis Associates, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Women Partners in Health, Austin, Texas
  - Willowbend Health & Wellness Associates, Plano, Texas
  - Medical Associates Inc., Menomonee Falls, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Proellex: Proellex 25 or 50 mg once daily
  One capsule Proellex 25 mg or 50 mg administered as daily oral doses for four (4) consecutive months during each treatment cycle
Period: Overall Study
Arm/Group | Proellex
Started | 175
Completed | 0
Not Completed | 175
Not completed — Study prematurely terminated | 175

BASELINE CHARACTERISTICS:
Population: Study prematurely terminated
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg Proellex | Proellex 50 mg | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Safety of Proellex Administered Once Daily for Three Treatment Cycles (4 Months Each Cycle)
Time Frame: 12 months
Population: Study prematurely terminated
Arm/Group | 25 mg Proellex | Proellex 50 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: No adverse events data is available.
Arm/Group | 25 mg Proellex | Proellex 50 mg
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated for safety reasons (Proellex studies were put on clinical hold due to liver toxicity). Sponsor was unable to pay vendor, and was therefore not provided with any study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights